CLINICAL TRIAL: NCT01492257
Title: Shared Decision Making in Patients With Osteoarthritis of the Hip and Knee
Acronym: SDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Stanford University (Other); Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UCSFSDMv1
Record Dates: First submitted 2011-12-06; First posted 2011-12-14 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis
Keywords: shared decision making; decision aids; total joint arthroplasty; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SDM Control (No Intervention): The control arm will consist of usual care, patients will receive existing educational materials.
- SDM Intervention (Experimental): RCT intervention will include a package of decision and communication aids question-asking, and information recall. The intervention includes digital video discs and booklets produced by the Foundation for Informed Medical Decision Making and Health Dialog; a question-prompting phone call with a trained health coach; audio-recordings of the patient-surgeon consultation; and a copy of the surgeon's dictated note.
  Interventions: Other: Shared Decision Making Intervention

INTERVENTIONS:
Other: Shared Decision Making Intervention — Digital video discs and booklets produced by the Foundation for Informed Medical Decision Making and Health Dialog; a question-prompting phone call with a trained health coach; audio-recordings of the patient-surgeon consultation; and a copy of the surgeon's dictated note.
  Arms: SDM Intervention

SUMMARY:
Total joint arthroplasty (TJA) is an effective procedure for reducing pain and improving function in patients with disabling osteoarthritis (OA) of the hip or knee. However, as with all invasive procedures, TJA is associated with certain risks and substantial costs. Since the indications for TJA are heavily dependent on patients' quality of life and expectations. TJA utilization rates vary widely throughout the United States, as seen with other 'preference-sensitive' procedures. Early evidence suggests shared decision making (SDM) strategies are effective in enhancing patient decision quality, or the degree to which treatment decisions reflect the preferences of fully informed patients, especially for preference-sensitive procedures like TJA. Despite these advantages, however, SDM has not been embraced or widely adopted in orthopaedics. To investigate this limited uptake, the investigators propose a series of evaluations of individual-level strategies. The investigators innovative and unique contribution is to approach patients, surgeons and healthcare purchasers as having symmetric and equally valid concerns about the benefits and cost associated with SDM. The investigators overall objective is to facilitate wider dissemination of SDM strategies in orthopaedic practices. The specific aims of the project are to assess, for SDM strategies, the impact on key patient, surgeon, and healthcare purchaser priorities; By achieving this aim our project will produce new interventions and incentives for disseminating SDM that are endorsed as feasible and acceptable by a coalition of patients, surgeons, and purchasers. The investigators plans for evaluation include a randomized controlled trial to evaluate the impact of SDM on outcomes of interest to patients, surgeons, and purchasers.

DETAILED DESCRIPTION:
We propose an RCT based on a non-randomized pilot study conducted at UCSF that included 115 patients who were referred for evaluation of hip and knee OA. The results of this pilot study suggested that DESI's were associated with greater patient knowledge, higher decision quality, higher patient and surgeon satisfaction, and no substantial impact on length of office visit or treatment decision. As in the pilot study, the RCT intervention will include a package of decision and communication aids shown in prior studies to increase patient knowledge, question-asking, and information recall. The intervention includes digital video discs and booklets produced by the Foundation for Informed Medical Decision Making and Health Dialog; a question-prompting phone call with a trained health coach; audio-recordings of the patient-surgeon consultation; and a copy of the surgeon's dictated note. The control arm will consist of usual care. Our primary outcome is the proportion of patients who arrive at an informed decision during the first visit. This outcome is of interest to patients, surgeons and healthcare purchasers, all of whom value efficiency and quality in delivery of care. Our hypothesis is that a higher proportion of patients in the intervention group will arrive at an informed decision during the first visit, as a result of being more knowledgeable and prepared for their visit, thus conserving resources while advancing quality. Secondary outcomes of interest will include treatment decision (e.g., surgical vs. non-surgical); patient and provider satisfaction; length of office visits; and adherence to treatment recommendations.

We will assess whether patients are informed or not using a survey instrument testing 19 consensus "key facts" developed by FIMDM based on evidence and expert opinion. We will measure whether patients arrive at a decision using the Stage of Decision Making instrument. We will administer both instruments immediately after the patient's first consultation with their surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Chronic unilateral or bilateral osteoarthritis of the hip or knee
* At least 18 years of age
* Must be psychosocially, mentally, and physically able to fully complete the questionnaires
* No previous joint replacement surgery
* First time visit to surgeon

Exclusion Criteria:

* Prior history of joint replacement surgery, ipsilateral or contralateral hip/knee replacement
* Subjects whose primary diagnosis is not osteoarthritis
* Subjects who cannot speak or read English
* Subjects who are cognitively impaired
* Subjects who refuse to complete surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Stage of decision making | Participants will be followed for the duration of the clinic visit, expected to last up to 4 hours
  We will measure the proportion of patients who will arrive at a more informed decision during the clinic visit through surveys administered before the clinic visit and immediately after the clinic visit. We will ask patients before the clinic visit what treatment decision they are leaning towards, how far along they are with this decision. We will ask patients after the clinic visit, what treatment they want and how far along they are with the decision.
Knowledge Score | Participants will be followed for the duration of the clinic visit, expected to last up to 4 hours
  We will assess whether patients are informed or not using a survey instrument testing 19 consensus "key facts" developed by the Foundation for Informed Decision Making (FIMDM) based on evidence and expert opinion.

SECONDARY OUTCOMES:
Treatment Decision | Participants will be followed for the duration of the clinic visit, expected to last up to 4 hours
  Patients will be asked in a questionnaire what treatment decision (surgical vs. non surgical) they chose immediately after their clinic visit.
Patient and Surgeon Satisfaction | Participants will be followed for the duration of the clinic visit, expected to last up to 4 hours
  Patients will be asked in the questionnaire to rate on a scale of 0-10, with 0 being lowest satisfaction, and 10 being highest satisfaction, how satisfied they were with the consultation. Surgeons will be asked, to rate on a scale of 0-10, how appropriate the content of the patient's questions were, how appropriate the number of the patient's questions were, how satisfied the surgeon was with the efficiency of the consultation, and overall satisfaction of the visit. Both surveys will be administered immediately after the clinic visit.
Length of office visit | Participants will be followed for the duration of the clinic visit, expected to last up to 4 hours
  A research associate will measure and record the start and stop time of the entire visit and the start and stop time of the surgeon consultation.
Adherence to treatment recommendations | At least 6 Weeks
  We will measure adherence to treatment recommendations through a 6 week follow up questionnaire administered at least6 weeks after the date of patient's clinic visit or 6 weeks after the date of the patient's surgery, if they had surgery. The questionnaire will ask patients what treatment decision they decided on, to rate on a scale of 0-10 how often they participated in physical therapy if prescribed, rate on a scale of 0-10 how often they took medication if prescribed within the past 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Bozic, MD, MBA, Principal Investigator — University of California, San Francisco; Vanessa Chiu, MPH, Study Director — University of California, San Francisco
Locations (2):
- United States (2):
  - Stanford University, Redwood City, California
  - University of California, San Francisco, San Francisco, California